CLINICAL TRIAL: NCT05800912
Title: Physical Therapy Students' Reflective Thinking With Narrative Photography in Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1821073
Record Dates: First submitted 2023-03-11; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Students
Keywords: Physiotherapy; Education; Heart transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to group allocation. A blinded assessor collected all baseline and post-intervention measures and entered the data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative photography group (Experimental): Students in the NP group performed training activities on empathy and care for patients undergoing heart transplantation.
  Interventions: Other: Narrative photography
- Traditional learning group (Active Comparator): Students in the TL group performed a conventional intervention without real patients.
  Interventions: Other: Traditional learning

INTERVENTIONS:
Other: Narrative photography — Students were shown real-life written stories, audio, and videos using a private online platform. The training activity included four modules: i) heart transplantation waiting list; ii) life expectancy, fear of death, and organ rejection; iii) post-transplant physical and functional limitations; and iv) lack of knowledge of physical exercise patients can perform.
  The students were encouraged to think about how they would feel if they had undergone heart transplantation. Afterward, they had to communicate these feelings using up to three photographs and reflective explanatory text.
  Two weeks later, the students met a heart transplantation expert patient followed by an educator-guided debate. Students' images were shared and discussed. Moreover, students were encouraged to explain their feelings and their acquired skills (two hours).
  Arms: Narrative photography group
Other: Traditional learning — A participatory lecture was carried out, in which cardiac rehabilitation in heart transplantation patients was explained. Then, there was an educator-guided debate about protocols and actions (one hour).
  Second, the students autonomously prepared clinical cases on physical limitations, physical exercise, risk factors, and life after transplantation (two hours).
  Two weeks later, the clinical session was held among students (2 hours). They adopted the roles of physical therapists or transplant patients to work on: i) post-transplant physical and functional limitations; ii) lack of knowledge of the physical exercise the patient can perform; iii) control of cardiovascular risk factors; iv) life post-transplant.
  Arms: Traditional learning group

SUMMARY:
Physical therapy students must learn about heart transplantation, and must be able to communicate with patients using empathy and moral sensitivity. The aim of the study is to compare the narrative photography (NP) and traditional learning (TL) methods applied to heart transplantation physical therapy, as they relate to physical therapy students' knowledge, empathy, satisfaction, and moral sensitivity.

DETAILED DESCRIPTION:
Physical therapy students must learn about heart transplantation. They need to know how to attend to the needs and emotions of these patients using empathy and moral sensitivity. The aim of the study is to compare the narrative photography (NP) and traditional learning (TL) methods applied to heart transplantation physical therapy, as they relate to physical therapy students' knowledge, empathy, satisfaction, and moral sensitivity.

This is a randomized contorlled trial with 117 participants of third year of Physiotherapy Degree. Students were divided into two groups: i) NP group (n = 56), and ii) TL group (n = 61).

Physical therapy knowledge in heart transplantation, empathy, and moral sensitivity were measured pre-intervention and post-intervention in both groups. Satisfaction was measured post-intervention in the NP group.

ELIGIBILITY:
Inclusion Criteria:

* Third-year physical therapy students who were studying the heart transplantation physical therapy course in a Physical therapy Degree.

Exclusion Criteria:

* Who did not meet the above inclusion criteria.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of physical therapy in heart transplantation | Baseline
  Knowledge of physical therapy in heart transplantation was measured using an ad-hoc multiple-choice questionnaire. To avoid any test preparation, students were not informed that there would be knowledge tests. The tests included 10 multiple-choice questions that assessed physical therapy knowledge of heart transplantation-related issues-this included rate of perceived exertion, cardiopulmonary exercise test, cardiac rehabilitation, symptoms, and signs. The minimum and maximum values were 0 and 10, respectively. Higher scores mean a better outcome.
Knowledge of physical therapy in heart transplantation | After the intervention (2 weeks)
  Knowledge of physical therapy in heart transplantation was measured using an ad-hoc multiple-choice questionnaire. To avoid any test preparation, students were not informed that there would be knowledge tests. The tests included 10 multiple-choice questions that assessed physical therapy knowledge of heart transplantation-related issues-this included rate of perceived exertion, cardiopulmonary exercise test, cardiac rehabilitation, symptoms, and signs. The minimum and maximum values were 0 and 10, respectively. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Empathy using the Interpersonal Reactivity Index | Baseline
  Empathy was measured using the Interpersonal Reactivity Index (IRI). The tool comprises 28 Likert questions ranging from 1 to 5 (1 = it does not describe me at all; 5 = it describes me very well). Four dimensions were explored using this questionnaire. These were perspective taking, fantasy, empathetic concern, and personal distress. Each scale score was the sum of the responses given for each item. The minimum and maximum values were 28 and 140, respectively. Higher scores reflected greater empathy.
Empathy using the Interpersonal Reactivity Index | After the intervention (2 weeks)
  Empathy was measured using the Interpersonal Reactivity Index (IRI). The tool comprises 28 Likert questions ranging from 1 to 5 (1 = it does not describe me at all; 5 = it describes me very well). Four dimensions were explored using this questionnaire. These were perspective taking, fantasy, empathetic concern, and personal distress. Each scale score was the sum of the responses given for each item. The minimum and maximum values were 28 and 140, respectively. Higher scores reflected greater empathy.
Moral sensitivity with the Revised Moral Sensitivity Questionnaire | Baseline
  Moral sensitivity was measured with the Revised Moral Sensitivity Questionnaire (RMSQ). The questionnaire included nine items rated on a 6-point Likert scale (1 = totally disagree, 6 = totally agree). The RMSQ comprises three dimensions. These are a sense of moral burden, moral strength, and moral responsibility. The minimum and maximum values were 9 and 54, respectively. Higher scores reflected greater moral sensitivity.
Moral sensitivity with the Revised Moral Sensitivity Questionnaire | After the intervention (2 weeks)
  Moral sensitivity was measured with the Revised Moral Sensitivity Questionnaire (RMSQ). The questionnaire included nine items rated on a 6-point Likert scale (1 = totally disagree, 6 = totally agree). The RMSQ comprises three dimensions. These are a sense of moral burden, moral strength, and moral responsibility. The minimum and maximum values were 9 and 54, respectively. Higher scores reflected greater moral sensitivity.
Satisfaction questionnaire | After the intervention (2 weeks)
  Satisfaction questionnaire was measured using a narrative photography questionnaire. This tool has previously been used to evaluate students' satisfaction with the narrative photography methodology as a tool to improve their skills and attitudes. This 32-item questionnaire was composed of sociodemographic questions, satisfaction with improving attitude, satisfaction with improving skills, and general satisfaction. It uses a 5-point Likert scale (1 = totally agree, 5 = totally disagree). The percentage of people who have rated each item is then calculated. Additionally, the questionnaire included a reflective open-ended question.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marqués Sulé, PhD, Principal Investigator — Univeristy of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leyva-Moral JM, Aguayo-Gonzalez M, Folch C, San Rafael S, Gomez-Ibanez R. Nursing students' perceptions of the efficacy of narrative photography as a learning method: A cross-sectional study. Nurs Health Sci. 2022 Jun;24(2):380-386. doi: 10.1111/nhs.12932. Epub 2022 Mar 3. PMID 35199453
- [Background] Leyva-Moral JM, Gomez-Ibanez R, San Rafael S, Guevara-Vasquez G, Aguayo-Gonzalez M. Nursing students' satisfaction with narrative photography as a method to develop empathy towards people with Hiv: A mixed-design study. Nurse Educ Today. 2021 Jan;96:104646. doi: 10.1016/j.nedt.2020.104646. Epub 2020 Nov 1. PMID 33160157